CLINICAL TRIAL: NCT00591604
Title: Use of High-Dose Vitamin D to Treat Vitamin D Deficiency Following Severe Burn Injury in Children I: A Pilot Study
Brief Title: High-Dose Vitamin D Deficiency in Burn Injury
Acronym: VitaminD
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: hurricane caused closure of hospital with PI not associated with Shriners Hospital for children
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-250
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Burn
Keywords: burn; vitamin D; nutrition; burn recovery
MeSH Terms: conditions — Burns | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Vitamin D administration
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Vitamin D, 50,000IU,once weekly for 8 weeks, then every other week for 4 weeks

SUMMARY:
High dose Vitamin D (50,000IU) therapy may increase bone mineral density/bone mineral content after large burns.

ELIGIBILITY:
Inclusion Criteria:

* 5+ yrs
* Burn size 40% or greater
* Patient can remain around Shriner Hospital for Children area for 16 weeks
* Agree to take Vitamin D

Exclusion Criteria:

* Age less than 5yrs
* Burn size less than 40%
* Pre-existing bone disease or healing fractures
* Underlying chronic disease-endocrine or cancer
* Kidney failure

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Increase in overall bone health | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David N Herndon, MD, Principal Investigator — University of Texas